CLINICAL TRIAL: NCT02912026
Title: An Open-Label, Single-Dose, Single-Period Study Designed to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]-F901318 Administered Via the Intravenous and Oral Routes to Healthy Male Subjects
Brief Title: Radiolabelled IV and Oral Metabolism Study of F901318
Acronym: ADME
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Major change to study design
Sponsor: F2G Biotech GmbH (Industry)
Collaborators: Quotient Clinical (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: F901318-01-08-16
Record Dates: First submitted 2016-09-21; First posted 2016-09-23 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2018-07

CONDITIONS: Invasive Aspergillosis
MeSH Terms: interventions — olorofim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous (Experimental): Intravenous AUC0-infinity
  Interventions: Drug: IV F901318
- Oral (Experimental): Oral AUC0-infinity
  Interventions: Drug: Oral F901318

INTERVENTIONS:
Drug: IV F901318 — Metabolic profile AUC 0 to infinity
  Arms: Intravenous
Drug: Oral F901318 — Metabolic profile AUC 0 to infinity
  Arms: Oral

SUMMARY:
Open label radiolabelled metabolism study of intravenous and oral solution forms of F901318. Five healthy male subjects will receive IV and five will receive an oral solution. Blood, urine and faeces will be collected over a period adequate to obtain 90% recovery of parent compound and to determine the metabolic profile of both IV and oral forms.

DETAILED DESCRIPTION:
Subjects will be screened for eligibility to participate in the study up to 28 days before dosing. Eligible subjects will be admitted to the clinical unit on the evening of Day -1 prior to investigational medicinal product (IMP) administration, and will be dosed on the morning of Day 1. In Cohort 1 (Regimen A), subjects will be dosed after a light breakfast; to assess tolerability of the IV administration, the first subject will be dosed at least 30 min prior to dosing the second subject. All subsequent dosing of the IV formulation will be staggered by at least 15 min. In Cohort 2 (Regimen B), subjects will be dosed following an overnight fast with an appropriate interval between subjects based on logistical requirements. Subjects will remain resident in the clinic up to 336 h post-dose (Day 15). It is planned that subjects will return to the clinical unit for 2 further 24 h residency periods on Day 21 and Day 28 if discharge criteria outlined in this protocol are not met. It is planned that subjects will be released from the study as a group when all subjects have achieved a mass balance cumulative recovery of >90% or <1% of the dose administered has been collected in urine and faeces within 2 separate, consecutive 24 h periods. If this occurs earlier than Day 28, collection of all samples (blood, urine and faeces) will be stopped and the subjects will undergo discharge assessments. If this criterion has not been met by all subjects following the Day 28 return visit, home collections of urine and faeces may be requested at the discretion of the investigator for individual subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males who do not wish to father children within the 6 months following IMP administration.
2. Age 40 to 65 years of age at the time of signing the ICF.
3. Body mass index of 18.0 to 35.0 kg/m2, with a weight of 50 to 100 kg.
4. Must be willing and able to communicate and participate in the whole study.
5. Subjects must be in good health as determined by a medical history, physical examination, 12-lead ECG and clinical laboratory evaluations.
6. Must have regular bowel movements (ie, average stool production of ≥1 and ≤3 stools per day).
7. Must provide written informed consent and agree to abide by the study restrictions
8. Must agree to use an adequate method of contraception during the study and for 6 months after study discharge

Exclusion Criteria:

1. Subjects who have received any IMP in a clinical research study within the previous 3 months prior to dosing.
2. Subjects who are study site employees, or immediate family members of a study site or sponsor employee.
3. Subjects who have previously been enrolled in this study or have previously been exposed to F901318.
4. History of any drug or alcohol abuse in the past 2 years.
5. Regular alcohol consumption in males >21 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine).
6. Current smokers and those who have smoked or used nicotine containing products (eg electronic cigarettes) within the last 6 months. A confirmed positive urine cotinine test at screening or admission.
7. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study.
8. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening.

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Mass balance | 28 days
  Metabolic profiling over 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Clinical, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No